CLINICAL TRIAL: NCT02385617
Title: Food Intake and Gut Hormone Release in Patients in Cancer Remission Who Have Undergone Upper Gastrointestinal Surgery
Brief Title: Food Intake and Gut Hormones in Patients Who Have Undergone Upper Gastrointestinal Surgery for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: University College Dublin (Other); University of Dublin, Trinity College (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRFSJ 0026; REC 2011/27/01 (Other: St. James's Hospital Research Ethics Committee)
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition
Keywords: Glucagon-Like Peptide 1; Peptide YY; Ghrelin; Satiety Response; Appetite; Hunger; Somatostatin; Octreotide; Anastomosis, Roux-en-Y; Digestive System Surgical Procedures; Pharmacologic Actions; Physiological Effects of Drugs; Endocrine System Diseases; Enteroendocrine Cells; Gastrointestinal Agents
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition; Endocrine System Diseases | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Esophagectomy (Experimental): Double blind single dose placebo-octreotide crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Total gastrectomy (Experimental): Double blind single dose placebo-octreotide crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Control - no surgery (Active Comparator): Double blind single dose placebo-octreotide crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Pancreaticoduodenectomy (Experimental): Double blind single dose placebo-octreotide crossover
  Interventions: Drug: Octreotide; Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Octreotide 100mcg (1mL) single dose, subcutaneously, into the lower abdomen, 50 minutes prior to eating
  Other Names: Sandostatin
Drug: Placebo — 0.9% saline (1mL) single dose, subcutaneously, into the lower abdomen, 50 minutes prior to eating

SUMMARY:
Improvements to treatment strategies for patients upper gastrointestinal cancers have produced an increasing population of people who remain free from disease recurrence in the long term. Weight loss and nutritional problems are common among patients who attain long-term remission and cure after surgery for upper gastrointestinal cancers. However, the mechanisms underlying these problems are not well understood. In this study the investigators aim to determine whether reduced food intake after upper gastrointestinal surgery is caused by early satiety related to exaggerated post-prandial gut hormone responses.

This is a randomized, double-blind, placebo controlled, crossover study of the effect of 100μg octreotide SC on ad libitum food intake in patients free from complications or recurrence at least one year post-oesophagectomy, gastrectomy or pancreaticoduodenectomy. A comparator group of age, weight and gender matched subjects will be studied concurrently, and caloric intake and subjective symptom scores after administration of octreotide versus placebo among surgical and comparator subjects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical procedure: Two-stage, three-stage or transhiatal oesophagectomy with gastric conduit reconstruction and pyloroplasty, total gastrectomy with Roux-en-Y reconstruction, pancreaticodueodenectomy, or matched unoperated healthy controls
2. At least one year in remission post-resection (surgical groups)

Exclusion Criteria:

1. Pregnancy, breastfeeding
2. Significant and persistent chemoradiotherapy and/or surgical complication
3. Other previous upper gastrointestinal surgery
4. Significant dysphagia or odynophagia, unable to eat
5. Other disease or medications which may affect satiety gut hormone responses
6. Active and significant psychiatric illness including substance misuse
7. Cognitive or communication issues or any factors affecting capacity to consent to participation
8. History of significant food allergy, certain dietary restrictions
9. Confirmed or suspected residual or recurrent disease after surgery, second primary malignancy
10. Other reconstruction (eg colonic or jejunal interposition)
11. Any contraindication to octreotide administration

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum calorie intake | 1 hour
  Total kcals consumed

SECONDARY OUTCOMES:
Post-prandial satiety gut hormone response | 2 hours
  GLP-1, PYY, OXM plasma concentrations
Subjective symptom scores | 3 hours
  Modified visual analogue scale scores

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MCh, FRCS, Principal Investigator — Department of Surgery, St. James's Hospital
Locations (2):
- Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin, Ireland
- Gastrosurgical Laboratory, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Background] le Roux CW, Welbourn R, Werling M, Osborne A, Kokkinos A, Laurenius A, Lonroth H, Fandriks L, Ghatei MA, Bloom SR, Olbers T. Gut hormones as mediators of appetite and weight loss after Roux-en-Y gastric bypass. Ann Surg. 2007 Nov;246(5):780-5. doi: 10.1097/SLA.0b013e3180caa3e3. PMID 17968169
- [Background] Martin L, Lagergren J, Lindblad M, Rouvelas I, Lagergren P. Malnutrition after oesophageal cancer surgery in Sweden. Br J Surg. 2007 Dec;94(12):1496-500. doi: 10.1002/bjs.5881. PMID 17668914
- [Background] Haverkort EB, Binnekade JM, de Haan RJ, Busch OR, van Berge Henegouwen MI, Gouma DJ. Suboptimal intake of nutrients after esophagectomy with gastric tube reconstruction. J Acad Nutr Diet. 2012 Jul;112(7):1080-7. doi: 10.1016/j.jand.2012.03.032. PMID 22889637
- [Background] Donohoe CL, McGillycuddy E, Reynolds JV. Long-term health-related quality of life for disease-free esophageal cancer patients. World J Surg. 2011 Aug;35(8):1853-60. doi: 10.1007/s00268-011-1123-6. PMID 21553202
- [Background] Reynolds JV, McLaughlin R, Moore J, Rowley S, Ravi N, Byrne PJ. Prospective evaluation of quality of life in patients with localized oesophageal cancer treated by multimodality therapy or surgery alone. Br J Surg. 2006 Sep;93(9):1084-90. doi: 10.1002/bjs.5373. PMID 16779881
- [Background] Miholic J, Orskov C, Holst JJ, Kotzerke J, Pichlmayr R. Postprandial release of glucagon-like peptide-1, pancreatic glucagon, and insulin after esophageal resection. Digestion. 1993;54(2):73-8. doi: 10.1159/000201016. PMID 8319842
- [Background] Miras AD, le Roux CW. Mechanisms underlying weight loss after bariatric surgery. Nat Rev Gastroenterol Hepatol. 2013 Oct;10(10):575-84. doi: 10.1038/nrgastro.2013.119. Epub 2013 Jul 9. PMID 23835488
- [Background] Koizumi M, Hosoya Y, Dezaki K, Yada T, Hosoda H, Kangawa K, Nagai H, Lefor AT, Sata N, Yasuda Y. Postoperative weight loss does not resolve after esophagectomy despite normal serum ghrelin levels. Ann Thorac Surg. 2011 Apr;91(4):1032-7. doi: 10.1016/j.athoracsur.2010.11.072. PMID 21440118
- [Background] Doki Y, Takachi K, Ishikawa O, Miyashiro I, Sasaki Y, Ohigashi H, Nakajima H, Hosoda H, Kangawa K, Sasakuma F, Motoori M, Imaoka S. Ghrelin reduction after esophageal substitution and its correlation to postoperative body weight loss in esophageal cancer patients. Surgery. 2006 Jun;139(6):797-805. doi: 10.1016/j.surg.2005.11.015. PMID 16782437
- [Background] Miyazaki T, Tanaka N, Hirai H, Yokobori T, Sano A, Sakai M, Inose T, Sohda M, Nakajima M, Fukuchi M, Kato H, Kuwano H. Ghrelin level and body weight loss after esophagectomy for esophageal cancer. J Surg Res. 2012 Jul;176(1):74-8. doi: 10.1016/j.jss.2011.09.016. Epub 2011 Oct 3. PMID 22137988
- [Result] Elliott JA, Jackson S, King S, McHugh R, Docherty NG, Reynolds JV, le Roux CW. Gut Hormone Suppression Increases Food Intake After Esophagectomy With Gastric Conduit Reconstruction. Ann Surg. 2015 Nov;262(5):824-29; discussion 829-30. doi: 10.1097/SLA.0000000000001465. PMID 26583672
- See also: Wellcome Trust-HRB Clinical Research Facility — http://www.sjhcrf.ie/
- See also: St James's Hospital, Dublin — http://www.stjames.ie/
- See also: University of Gothenburg — http://www.gu.se/english